CLINICAL TRIAL: NCT06695143
Title: Antimicrobial Adjuvants to Revert the Imbalance of Skin Microbiota for Improved Outcomes of Complicated Cutaneous Leishmaniasis Treatment in Ethiopia
Acronym: AIM-CL
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Armauer Hansen Research Institute (AHRI), Ethiopia (Unknown); Arba Minch University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIM-CL
Record Dates: First submitted 2024-11-08; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: Cutaneous Leishmania; Complicated cutaneous leishmania
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Fusidic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment - SoC + fusidic acid 2% cream (Experimental): 4 weeks SSG (SoC) with 2 weeks twice daily topical application of fusidic acid 2% cream
  Interventions: Drug: Fusidic Acid
- Vehicle - SoC + vehicle cream (Active Comparator): 4 weeks SSG (SoC) with 2 weeks twice daily topical application of vehicle cream
  Interventions: Other: Vehicle cream
- Control - SoC (No Intervention): 4 weeks SSG (SoC) only

INTERVENTIONS:
Drug: Fusidic Acid — Fusidic acid 2% cream
  Arms: Treatment - SoC + fusidic acid 2% cream
Other: Vehicle cream — Cetomacrogol cream
  Arms: Vehicle - SoC + vehicle cream

SUMMARY:
This clinical trial aims to evaluate the effectiveness of combining the standard treatment for complicated cutaneous leishmaniasis (CL), sodium stibogluconate (SSG), with either topical fusidic acid 2% cream or a vehicle cream without active ingredient. The goal is to assess whether this combination improves treatment outcomes by restoring the balance of the skin microbiome (dysbiosis) in patients with severe CL, a condition common in Ethiopia.

The study will compare three treatment groups:

* Fusidic Acid Group: SSG plus topical fusidic acid for 2 weeks.
* Vehicle Cream Group: SSG plus topical vehicle cream for 2 weeks.
* Control Group: SSG only, with no topical treatment.

The primary objective is to determine if the addition of fusidic acid improves treatment outcomes compared to SSG alone, as measured by substantial improvement in the index lesion at the end of treatment (EoT).

A total of 180 patients will be enrolled at two hospitals in Ethiopia. The trial will run for 24 months, with a focus on understanding how restoring the skin microbiome can improve CL treatment outcomes and potentially provide a low-cost, accessible treatment strategy for CL patients.

ELIGIBILITY:
Clinically suspected complicated CL patients visiting the study site meeting the following inclusion criteria and none of the exclusion criteria:

Inclusion:

* Clinical diagnosis of CL
* Need for systemic treatment (1 or more of these criteria)

  * Mucosal involvement of lesion or at risk for mucosal involvement (< 1 cm from the nose, eyes and vermillion border of the lips)
  * Lesion size >4 cm
  * >4 lesions
  * Lesions on joints or fingers
  * Lesions previously not responding to local treatment
  * Lesions unsuitable for local treatment (e.g., eyelids)
  * Lesions with signs of dissemination (satellite lesions, nodular lymphangitis, sporotrichoid pattern)
* Age > 4 (minimum age to receive systemic treatment with SSG)
* At least one lesion eligible for treatment* (meeting all criteria below)

  * lesion with surface change, including ulcerated, crusted and scaly lesions
  * distinguishable from other lesions (minimum 0.5 cm apart)
  * no mucosal involvement against which a topical agent would likely not be effective (e.g., lesions that are located too deep within the nasal passages or on the inner lip, where proper application is challenging and the ointment may be easily removed or not adequately absorbed)
* Willing and able to provide informed consent. For participants under the age of 18, parental or caregiver consent is required. Additionally, assent must be obtained from adolescents aged 12 to 17
* Willing to be hospitalized for 4 weeks

Exclusion:

* DCL patients
* Only lesions not eligible for treatment*
* Currently on treatment or having received non-traditional antileishmanial treatment (cryotherapy, thermotherapy, sodium stibogluconate, meglumine antimoniate, paromomycin, pentamidine, AmBisome, miltefosine, non-liposomal amphotericin B) in the past 1 month
* Currently on or having received topical antibiotic treatment for CL lesion(s) in the past 1 month
* Currently on or having received systemic antibiotic treatment in general in the past 1 month
* Currently in need for systemic antibiotics
* Pregnant (positive pregnancy test at D0) or breastfeeding
* Abnormal lab values

  * Hemoglobin < 5.0g/100mL
  * Platelets < 50 x 10^9/L
  * White blood count < 1 x 10^9/L
  * ASAT/ALAT > 3x upper normal range
  * Creatinine above the normal limit
* Prolonged QTc interval or arrythmia on ECG or history of arrythmias
* Known serious kidney or liver disease
* Known allergies to one of the study components/medications
* Serious adverse reaction to a previous SSG dose *If a patient has multiple lesions, of which some are eligible for treatment and others are not, the patient can still be involved in the study. Only the eligible lesions will be subjected to treatment and outcome assessment.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Improvement of index lesion at EoT | 28 days
  To assess if 4 weeks SoC with 2 weeks application of 2% fusidic acid twice per day (Arm 1, Treatment) is superior to 4 weeks SoC only (Arm 3, Control) for complicated CL patients, in terms of reaching at least substantial improvement* of the index lesion** at the end of treatment (EoT).
  *Substantial improvement is defined as >50% flattening and >50% re-epithelization compared to the baseline assessment. Improvement will be measured for each lesion. At least the index lesion needs to be improved or cured for a patient to be considered substantially improved.
  **Index lesion is defined as the largest lesion eligible for treatment.

SECONDARY OUTCOMES:
Arm 1 superiority to arm 3 - index lesion | 42 days
  To assess if Arm 1 is superior to Arm 3, using an ordinal (no improvement, minor improvement, substantial improvement, cure, relapse) and continuous (% re-epithelization/flattening) outcome measures for the index lesion at EoT and D42
Arm 1 superiority to arm 3 - lesions eligible for treatment | 42 days
  To assess if Arm 1 is superior to Arm 3, using binary (at least substantial improvement), ordinal (no improvement, minor improvement, substantial improvement, cure, relapse) and continuous (% re-epithelization/flattening) outcome measures for all lesions eligible for treatment individually and combined at EoT and D42
Proportion of participants that reach substiantial improvement - arm 1 vs arm 2 | 42 days
  To compare the proportion of patients that reach at least substantial improvement of the index lesion, all lesions combined and individually at EoT and D42 between patients who received SoC with topical 2% fusidic acid (Arm 1, Treatment), and those who received SoC combined with topical vehicle cream (Arm 2, Vehicle)
Proportion of participants that reach substiantial improvement - arm 2 vs arm 3 | 42 days
  To compare the proportion of patients that reach at least substantial improvement of the index lesion, all lesions combined and individually at EoT and D42 between patients who received SoC combined with topical vehicle cream (Arm 2, Vehicle), and those who received SoC only (Arm 3, Control)
Cycles needed for final cure | 180 days
  To compare the number of cycles needed to reach final cure per treatment arm
Proportion of cured patients at day 180 | 180 days
  To determine the proportion with 95% CI of patients that reach cure without relapsed or worsening at day 180 for the three treatment arms
Quality of life - patient reported outcome | 180 days
  To compare change over time of patient-reported outcomes - the dermatological life quality index (DLQI) scores and global assessment - per treatment arm
Safety and acceptability | 180 days
  To assess safety and acceptability of treatment arms
  a) Withdrawal from study intervention: proportion and 95% CI of patients withdrawn from intervention, per arm b) Adverse events: number and proportion of patients with adverse events, per arm c) Cumulative incidence of adverse events (AEs) related to the study drug d) Recommendability: acceptability and recommendability score (0-10) given by patients after treatment completion, per arm
Stability microbial diversity | 180 days
  To determine the stability of microbial diversity in the healthy skin over time
Increase microbial diversity | 180 days
  To assess the increase in microbial diversity indices within each trial arm at D14, EoT, D42 and M6 compared to D0.
Correlation microbial diversity and substantial improvement | 180 days
  To determine whether increase in microbial diversity at EoT compared to D0 is correlated with substantial improvement of the index lesion and all lesions combined at EoT for the three trial arms
Correlation microbial diversity and cure without relapse | 180 days
  To determine whether increase in microbial diversity at M6 compared to D0 is correlated with cure without relapse at M6, for the three trial arms

CONTACTS AND LOCATIONS:
Overall Officials: Johan Van Griensven, Prof, Principal Investigator — Head of department of clinical sciences
Locations (2):
- Ethiopia (2):
  - Arba Minch General Hospital, Arba Minch
  - Chencha Primary Hospital, Chencha

IPD SHARING:
Plan to Share IPD: No